CLINICAL TRIAL: NCT03575858
Title: Comparison of Barrel Shaped and Tapered Interdental Brushes in the Management of Peri-implant Mucositis and Gingivitis in Healthy Individuals: A Randomized Controlled Single Blinded Clinical Trial
Brief Title: The Effect of Different Shapes of Interdental Brushes in the Management of Peri-implant Mucositis and Gingivitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Barrel shaped interdental brush went out of production
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jia Hui Fu, Assistant Professor, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/01230
Record Dates: First submitted 2018-06-06; First posted 2018-07-03 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Dental Implants, Single-Tooth
Keywords: Single dental implants; Barrel Shaped Interdental toothbrush; Tapered Interdental toothbrush; peri-implant mucositis and gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into the barrel shaped (test) and tapered (control) interdental brushes groups
Who Masked: Outcomes Assessor
Masking Description: The study examiner who will be doing the clinical examination and collecting the study data will be blinded to the group allocation; however it is not possible to blind the study subjects to the group allocation. The clinician, who will be performing the treatment and providing oral hygiene instructions, will open the envelope containing the subject's group allocation after non-surgical periodontal therapy but before giving the oral hygiene instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barrel shaped interdental brushes (Experimental): test group
  Interventions: Device: Barrel shaped interdental brush
- Tapered interdental brushes (Active Comparator): control group
  Interventions: Device: Tapered interdental brush

INTERVENTIONS:
Device: Barrel shaped interdental brush — Barrel shaped interdental brush Size SS 0.8mm
  Arms: Barrel shaped interdental brushes
Device: Tapered interdental brush — Tapered interdental brush Size SS 0.6mm
  Arms: Tapered interdental brushes

SUMMARY:
Rehabilitation of edentulous spaces with dental implants has become a routine treatment option as implants enjoy high survival rates over time. Accompanying this increase in implant use, epidemiological studies have also reported escalating incidences of peri-implant diseases. A recent meta-analysis reported that peri-implant mucositis and peri-implantitis had high estimated weighted mean prevalences of 43% and 22% respectively. It is common knowledge that gingivitis is the precursor of periodontitis. Similarly, peri-implant mucositis too precedes peri-implantitis, which is a very challenging condition to treat. Therefore, it is strongly recommended that peri-implant mucositis is managed effectively and in a timely manner.

In order to reduce the inflammatory burden within the periodontium, mechanical plaque removal is of utmost importance. Mechanical debridement alone, without any adjunctive aids e.g. chlorhexidine, was found to be effective in preventing per-implant mucositis in short-term clinical trials but did not always result in complete resolution of inflammation (Heitz-Mayfield, et al. 2011, Schwarz, et al. 2015). Therefore, it can be speculated that patient administered home care may play a role in eliminating soft tissue inflammation over time.

The study aims to investigate and compare the efficacy of the barrel shaped and tapered interdental brushes in reduction of soft tissue inflammation through removal of interproximal plaque at both tooth and implant sites in patients with moderately rough surface tissue level or bone level dental implants, which were restored with single screw or cement retained crowns and in function for the past 2- 5 years.

The hypothesis of the study is that The barrel shaped interdental brush can remove more supra- and sub-gingival plaque and thus have more reduction in soft tissue inflammation, compared to the tapered interdental brush.

DETAILED DESCRIPTION:
There are two study phases during the whole course of the study.

1) Examiner Calibration: 15 volunteers will be recruited for examiner calibration before the study period. The intra-examiner reliability will be assessed using intraclass correlation coefficient. The following clinical parameters will be collected at day 0 and day 7.

Clinical Parameters:

i. Probing pocket depths (PPD) (6 points per tooth) ii. Full mouth bleeding score (FMBS) iii. Plaque at 8 sites (mesiobuccal, mesial, mesiolingual, lingual, distolingual, distal, distobuccal, and buccal) per implant

2) Study phase: Stratified randomized single-blinded clinical controlled trial with 2 parallel arms is designed to achieve the aims of this research project. Study participants who are visiting University Dental Cluster or any other dental clinics or hospitals will be referred for this study. They will be enrolled at NUH University Dental Cluster if they fulfill the study inclusion and exclusion criteria. They will be randomly assigned into the barrel shaped (test) and tapered (control) interdental brushes groups and reviewed at 2 weeks (± 3 days) and 4 weeks (± 3 days).

Randomization:

Study subjects will be randomly assigned to either test or control group based on a computer generated randomization code after the screening of inclusion and exclusion criteria and signing of the informed consent form.

Blinding and Allocation Concealment:

The study examiner who will be doing the clinical examination and collecting the study data will be blinded to the group allocation; however, it is not possible to blind the study subjects to the group allocation. The clinician, who will be performing the treatment and providing oral hygiene instructions, will be given a sequentially numbered envelope containing the subject's group allocation after non-surgical periodontal therapy has been performed and before giving the oral hygiene instructions.

i. Probing pocket depths (PPD) (6 points per tooth) ii. Full mouth bleeding score (FMBS) iii. Full mouth plaque score (FMPS) iv. Plaque at 8 sites (mesiobuccal, mesial, mesiolingual, lingual, distolingual, distal, distobuccal, and buccal) per implant v. Characteristics of the implant and implant crown: tissue level or bone level, supra- or submucosal margin, degree of overcontour as seen on periapical radiograph vi. Peri-apical radiograph of implant taken with parallel technique

Clinical parameters (i) to (iv) will be performed at baseline, 2-weeks and 4-weeks post instrumentation.

Clinical parameter (v) and (vi) will be performed at baseline.

Radiographic Analysis:

Peri-apical radiographs will be only taken with paralleling technique to determine that there is no peri-implant bone loss at baseline.

The sample size is calculated based on changes in mean bleeding on probing (BOP) (primary outcome measure) between baseline and at 2 weeks post instrumentation review. Based on a previous study (Larsen, et al. 2017), investigators calculated that 88 subjects (44 per group) would be needed with 5% significance level and 80% statistical power. If investigators expect an attrition rate of 20%, a total of 110 subjects (55 per group) will be needed.

Statistical Analysis:

Intention-to-treat analysis on the primary outcome variable (BOP) will be performed. Last-observation-carried-forward method will be used in the event of subjects lost to follow-up to the end of the study.

Descriptive statistics (mean and standard deviation for continuous variable; frequency and percentage for categorical variable) will be reported to summarize the baseline characteristics of study participants. Primary analysis will be patient-level analysis and secondary analysis will be implant-level analysis. One implant, will be randomly selected by computer generated random number, from each recruited subjects for patient-level analysis. All implants from the recruited subjects will be included in the implant-level analysis.

At patient-level analysis, to examine the effect of shape of interdental brush, difference-in-difference technique will be used for study the changes of outcomes (e.g. BOP, PPD, FMBS and FMPS) from baseline at 2-weeks. Two-way ANOVA test with adjusting for implant types will also be performed to study the effect of interdental brush shape in the form of changes in BOP, PPD, FMBS and FMPS, at 2-week. Similar analysis will be replicated for secondary study endpoint at 4-week. Generalized estimating equation (GEE) will be applied to incorporate repeated measures data collected at 2- and 4-weeks. Baseline data and types of implants will be adjusted in the model.

At implant-level analysis, to adjust for within-patient dependency, multilevel mixed effects model will be built to assess the effect of interdental brush shape on the study outcome variables (e.g. BOP, PPD, FMBS and FMPS) over time. A multilevel hierarchical three-level structure was chosen with three levels of analysis being: timing of follow-up measurements (level 1), implant (level 2), and patient (level 3). Baseline values of study outcome variables and types of implants will be adjusted in the model.

Significance level for all analysis is set at p-value <0.05. All statistical analysis will be carried out using STATA SE Version 15.0 (StataCorp. 2017. Stata Statistical Software: Release 15. College Station, TX: StataCorp LLC).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years old
* Medically healthy (ASA I or II)
* Baseline plaque score of at least 75%
* Probing depths of 4mm or less
* Presence of interdental spaces that will allow an interdental brush (Size SS 0.8mm for barrel-shaped interdental brush and 0.6mm tapered interdental brush) to pass through without soft tissue trauma
* Single moderately rough tissue level or bone level dental implants, which were restored with a single cement or screw-retained crown and in function for the past 2-5 years
* Implants should have peri-implant mucositis defined as bleeding on probing without peri-implant bone loss after physiological remodelling (Rosen, et al. 2013)
* Implants with at least 1mm of keratinized peri-implant mucosa

Exclusion Criteria:

* Embrasure space between the implant and adjacent tooth or between teeth is non-existent or too small to permit the use of an interdental brush
* Self-declared pregnancy
* Heavy smokers (1 pack a day)
* Uncontrolled or poorly controlled medical conditions e.g. diabetes (HBA1c 8.5% and above)
* Untreated oral conditions e.g. active periodontitis
* On medications that will cause gingival enlargement
* Any hyperplastic interdental papilla that will hinder interdental cleaning
* Antibiotics intake within the past 3 months
* Parkinson's disease and other debilitating diseases

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in peri-implant tissue health as assessed by bleeding on probing (BOP). | Baseline, 2-week and 4-week
  The changes in BOP at 6 sites per implant at 3 time points - from baseline to 2-weeks and to 4-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Hui Fu, Master, Principal Investigator — National University Health System, Singapore

IPD SHARING:
Plan to Share IPD: No